CLINICAL TRIAL: NCT00205426
Title: Natrecor® (Nesiritide) as a Nitric Oxide Sparing Agent in Patients Undergoing Lung Transplantation
Brief Title: Natrecor for Pulmonary Hypertension in Lung Transplants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-2005-0185
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary hypertension in lung transplant recipients
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Natrecor infusion (Experimental): Nesiritide
  Interventions: Drug: Natrecor

INTERVENTIONS:
Drug: Natrecor — Natrecor will be initiated as a bolus dose of 2 mcg/kg followed by a continuous infusion via infusion pump after induction of anesthesia but prior to incision. Natrecor infusion will be started at the recommended rate of 0.01mcg/kg/min. This dose may be adjusted by the investigator(s) only based on hemodynamic monitoring and pulmonary parameters. Study drug will be infused for a minimum of 24 hours and a maximum of 96 hours.
  Other Names: nesiritide

SUMMARY:
This study seeks to demonstrate that Natrecor® (nesiritide) is safe and effective and has a favorable hemodynamic profile in lung transplant recipients that will allow for the avoidance of inhaled nitric oxide (iNO) use. It is estimated that the use of nesiritide will decrease the otherwise historically mandated use of iNO by 50%, as compared to the necessity of iNO use by matched historical controls.

DETAILED DESCRIPTION:
A condition called ischemic reperfusion injury (IRI) occurs in all lung transplants. The amount of reperfusion injury varies from person to person. IRI occurs when the blood supply to tissue (in this case, transplanted lung(s)) is decreased and then is restored. IRI can cause a decrease in function in a newly transplanted lung. When this occurs, or when people have pulmonary hypertension (high blood pressure in your lungs), doctors use Nitric Oxide to improve the pressure and blood supply to the transplanted lung. Nitric Oxide (NO) is given by inhalation while patients are on a ventilator (breathing machine). Because NO must be given by a ventilator and because patients on ventilators must be in an intensive care unit, the cost of treating people with NO is very high. NO can also cause rebound pulmonary hypertension (high blood pressure in the lungs that reoccurs) when it is stopped. Because of these reasons, doctors are looking for other treatments for IRI and pulmonary hypertension. A drug called Natrecor has been shown to reduce pulmonary pressures in heart transplant patients. Doctors believe it may be helpful to lung transplant patients as well.

ELIGIBILITY:
Inclusion Criteria:

* Single or double lung transplant or heart/lung transplant recipient
* Planned use of Natrecor
* Pulmonary artery (PA) systolic pressures > 35

Exclusion Criteria:

* Previous lung transplant
* Use of Prolastin after pneumonectomy
* Mean arterial pressure of < 55
* Known allergy or sensitivity to nesiritide
* Females of childbearing potential with a positive pregnancy test or women who are breast feeding
* Use of nesiritide, for any reason, within 30 days prior to transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2005-08; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and efficacy of Natrecor® in reducing nitric oxide used perioperatively in patients undergoing single or double lung transplantation who have or are at risk for developing pulmonary hypertension

SECONDARY OUTCOMES:
To compare total cost-effective evaluation between patients receiving Natrecor and those who received iNO
To compare length of stay in the Intensive Care Unit (ICU)
To compare renal function as defined by peak serum creatinine and calculated creatinine clearance during the first 72 hours post-transplant
To compare necessity of CPB between Natrecor® versus nitric oxide
To compare hemodynamic parameters
To compare length of stay (total)
To compare time to dry weight
To compare duration of mechanical ventilation
To compare pulmonary parameters
To compare IRI via chest x-ray and PAO2/FIO2 ratio

CONTACTS AND LOCATIONS:
Overall Officials: Robert Love, MD, Principal Investigator — University of Wisconsin Medical School
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States